CLINICAL TRIAL: NCT00412607
Title: NaviStar ThermoCool Catheter for Endocardial RF Ablation in Patients With Ventricular Tachycardia
Brief Title: Catheter Evaluation for Endocardial Ablation in Patients With Ventricular Tachycardia
Acronym: VT-CoA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI40036
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia; Heart Diseases; Arrhythmia
MeSH Terms: conditions — Tachycardia, Ventricular; Heart Diseases; Arrhythmias, Cardiac

ARMS (1):
- NaviStar ThermoCool Catheter (Experimental)
  Interventions: Device: NAVISTAR® THERMOCOOL® Catheter

INTERVENTIONS:
Device: NAVISTAR® THERMOCOOL® Catheter — The primary objective is to provide additional, corroborative safety data for the NAVISTAR THERMOCOOL catheter for the treatment of subjects with sustained, monomorphic VT or incessant VT associated with coronary artery disease

SUMMARY:
The primary objective is to provide additional corroborative safety and efficacy data for the Navistar ThermoCool catheter for the treatment of subjects with ischemic Ventricular Tachycardia.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, single-arm, multi-center condition of approval evaluation. The device is currently FDA approved for commercial distribution. Subjects with ischemic ventricular tachycardia will be considered for the condition of approval study. This study will be conducted at up to 30 centers in a minimum of 249 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Documented spontaneous episodes of sustained ventricular tachycardia (must satisfy one)

   1. For patients with ICDs: Documented episodes must be four (4) or greater for entry into the study.
   2. For patients without ICDs: Documented episodes must be two (2) or greater within two (2) months and the assessment will be performed by a review of ECGs and hospitalization records.
   3. Incessant VT due to prior myocardial infarction (defined as present for more than one (1) hour and refractory to or immediately recurrent after administration of antiarrhythmic medication and cardioversion).
2. Spontaneous occurrence of symptomatic ventricular tachycardia despite antiarrhythmic drug therapy or ICD intervention.
3. Left ventricular ejection fraction > 10% as estimated by echocardiography, contrast ventriculography or radionuclide imaging within the previous ninety (90) days.
4. Age eighteen (18) years or older.
5. Signed Patient Informed consent form.
6. Able and willing to comply with all pre-, post-, and follow-up testing requirements.

Exclusion Criteria:

1. Definite protruding left ventricular thrombus on pre-ablation echocardiogram.
2. Myocardial infarction within the preceding two (2) months. Patients with incessant VT (defined as present for more than one (1) hour and refractory to or immediately recurrent after administration of antiarrhythmic medication and cardioversion) may be enrolled if their MI is at least three (3) weeks old.
3. Patients with idiopathic VT.
4. Other disease process likely to limit survival to less than twelve (12) months.
5. Class IV heart failure.
6. Serum creatinine of > 2.5 mg/dl.
7. Thrombocytopenia (defined as platelet count <80,000) or coagulopathy.
8. Contraindication to heparin.
9. Women who are pregnant.
10. Cardiac surgery (i.e. ventriculotomy, atriotomy) within the past two (2) months. Patients with incessant VT (present 50% of the time with intervention for a period >12 h) may be enrolled if their surgery is at least three (3) weeks old.
11. Acute illness or active systemic infection.
12. Unstable angina.
13. Severe aortic stenosis or flail mitral valve.
14. Uncontrolled heart failure.
15. Significant congenital anomaly or medical problem that, in the opinion of the Principal Investigator, would preclude enrollment in the study.
16. Enrolled in an investigational study evaluating another device or drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

REFERENCES:
- [Derived] Marchlinski FE, Haffajee CI, Beshai JF, Dickfeld TL, Gonzalez MD, Hsia HH, Schuger CD, Beckman KJ, Bogun FM, Pollak SJ, Bhandari AK. Long-Term Success of Irrigated Radiofrequency Catheter Ablation of Sustained Ventricular Tachycardia: Post-Approval THERMOCOOL VT Trial. J Am Coll Cardiol. 2016 Feb 16;67(6):674-683. doi: 10.1016/j.jacc.2015.11.041. PMID 26868693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on April 3, 2007. Subject enrollment was completed on May 19, 2009 after reaching the minimum enrollment criteria of two hundred forty-nine (249) subjects. Subject follow-up was completed on June 8, 2012.
Groups:
- NAVISTAR THERMOCOOL Catheter: NaviStar ThermoCool Deflectable Diagnostic/Ablation Catheter for the Treatment of Ventricular Tachycardia.
Period: Overall Study
Arm/Group | NAVISTAR THERMOCOOL Catheter
Started | 249
Started Study Catheter | 233
Completed | 145
Not Completed | 104
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 19
Not completed — Death | 61
Not completed — Not meet inclusion/exclusion Criteria | 15

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who signed the informed consent form and were eligible for inclusion in the clinical study
Arm/Group | NAVISTAR THERMOCOOL Catheter
Number analyzed (Participants) | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 234
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0
  Black | 14
  Caucasian | 229
  Hispanic | 4
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 249

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects That Expire From All-cause Mortality Within 12-months Post Ablation.
Description: The long-term primary safety endpoint is the percentage of subjects that expire from all-cause mortality within 12-months post ablation.
Time Frame: 12-month post ablation
Population: Safety analysis population - subjects who underwent insertion of the study catheter.
Measure: Number (95% Confidence Interval); unit: percentage of mortality
Arm/Group | NAVISTAR THERMOCOOL Catheter
Number analyzed (Participants) | 233
percentage of mortality | 13.3 [0 to 17.5]
Statistical Analysis 1: Comparison: NAVISTAR THERMOCOOL Catheter; Assumptions for sample size calculation: 10% attrition rate, Type I error of 0.05, anticipated 12-month mortality rate is 0.19, a region of indifference of 0.07, power of 0.8; the required sample size is 249 per nQuery Exact test for single proportion method. The null hypothesis is that the 12-month mortality rate is greater than or equal to 0.26; the alternative is that the rate is less than 0.26. This hypothesis is evaluated with one-sided exact binomial test at α= 0.05; Test type: Superiority or Other; Fisher Exact; Percentage of mortality = 13.3, 95% CI 1-sided [upper limit 17.5] — The 95% confidence interval is a one-sided with upper confidence level = 17.5% computed using the exact binomial test

2. Secondary Outcome: Percentage of Subjects Achieved Acute Success
Description: Acute success was defined as the subjects receiving successful ablation of all targeted Ventricular Tachycardia (VT) and no recurrence prior to hospital discharge.
Time Frame: Duration from post-procedure to hospital discharge, up to 2 days
Population: Subjects in the efficacy analysis cohort who had targeted ventricular tachycardia ablated were included. Efficacy Analysis Cohort includes subjects who are enrolled and treated with the study catheter in compliance with the protocol and treated specifically for the study-related arrhythmia.
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR THERMOCOOL Catheter
Number analyzed (Participants) | 215
Percentage of participants | 74.9

3. Primary Outcome: The Percentage of Subjects Who Experienced Cardiovascular-specific Adverse Events (CSAE) Within Seven Days of the Ablation Procedure.
Description: The acute primary safety endpoint is the percentage of subjects who experienced cardiovascular-specific adverse events (CSAE) within seven days of the ablation procedure.
Time Frame: Seven days post ablation procedure
Population: Safety Analysis Cohort - defined as subjects who underwent insertion of the study catheter.
Measure: Number (95% Confidence Interval); unit: percentage of Adverse Event
Arm/Group | NAVISTAR THERMOCOOL Catheter
Number analyzed (Participants) | 233
percentage of Adverse Event | 4.3 [0 to 7.2]

4. Secondary Outcome: Percentage of Subjects Who Achieved Chronic Effectiveness
Description: Chronic effectiveness is defined as subjects without recurrence of sustained monomorphic ventricular tachycardia (SMVT) at 6 month follow-up. For subjects with Implantable Cardioverter Defibrillator (ICD), recurrences of SMVT were defined as appropriate ICD shock therapies. For subjects without ICDs, recurrences of SMVT were recorded in the follow-up visits form. Besides SMVT, recurrence of incessant VT was also captured in this study. Recurrence of incessant VT was recorded up to 6 month post ablation procedure but not beyond.
Time Frame: 6-month follow up
Population: Subjects in the Efficacy analysis cohort who had available chronic effectiveness outcomes were included
Measure: Number; unit: Percentage of participants
Arm/Group | NAVISTAR THERMOCOOL Catheter
Number analyzed (Participants) | 184
Percentage of participants | 62.0

5. Secondary Outcome: Number of Subjects Achieved Long-term Efficacy Success
Description: Long-term success is defined as patient-reported non-recurrence of Ventricular Tachycardia (VT) at the12-month, second year, and third year phone follow-ups.
Time Frame: 3-year follow up
Population: Subjects in the efficacy analysis cohort who completed 12-month, 2-year, or 3-year follow-up and had available long-term efficacy outcomes at the corresponding time points were included.
Measure: Number; unit: participants
Groups:
- Total: Total number of subjects who completed 12-month, 2-year, and 3-year follow-up respectively.
- Reported Recurrence: Subjects reported recurrence of Ventricular Tachycardia (VT) at 12-month, 3-year follow-up visit
- Reported No Recurrence: Subjects reported no recurrence of Ventricular Tachycardia (VT) at 12-month, 3-year follow-up visit
Arm/Group | Total | Reported Recurrence | Reported No Recurrence
Number analyzed (Participants) | 176 | 176 | 176
participants
  12-Month Follow-up | 176 | 40 | 136
  2-Year Follow-up | 161 | 48 | 113
  3-Year Follow-up | 141 | 34 | 107

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction at 6 Month From Baseline
Description: Change in Left Ventricular Ejection Fraction (LVEF) from baseline to 6 month follow up. LVEF is a measure of the percentage of blood leaving heart each time it contracts. Baseline LVEF data were collected at pre ablation procedure, at hospital discharge, and at the 6-month follow-up visit.
Time Frame: 6-month follow up
Population: Efficacy analysis cohort subjects with LVEF data available. The statistics for Baseline and 6-month were based on data available from 219 and 166 subjects respectively; the mean change was based on 163 subjects with data at both Baseline and 6-month. Hence the mean change is not the simple subtraction between Baseline and 6-month.
Measure: Mean (Standard Deviation); unit: percentage of blood leaving the heart
Arm/Group | NAVISTAR THERMOCOOL Catheter
Number analyzed (Participants) | 219
percentage of blood leaving the heart
  Baseline (Pre-Ablation) | 30.6 (12.5)
  6-Month | 32.9 (11.53)
  Change from Baseline | 0.9 (8.23)

ADVERSE EVENTS:
Time Frame: 3-year follow up
Description: Serious adverse events (SAE) were those that meet the protocol definition of SAE, excluding the Cardiovascular Specific Adverse Events occurring within 7 days of the ablation procedure, but including deaths that occurred within the time frame. Deaths occurring after 7 days post-ablation were considered non-serious per the protocol definition.
Arm/Group | NAVISTAR THERMOCOOL Catheter
Serious Adverse Events (participants affected / at risk) | 37/233
Other Adverse Events (participants affected / at risk) | 177/233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVISTAR THERMOCOOL Catheter (N=233)
Bradycardia (Cardiac disorders) | 1 (1)
Death (Cardiac disorders) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 5 (5)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 3 (3)
Coronary Artery Disease Intervention (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 8 (8)
Pulseless Electrical Activity at Device Site (Cardiac disorders) | 1 (1)
Staphylococcus (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 1 (1)
MRSA (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection/Urinary Retention Retention (Infections and infestations) | 5 (6)
Fluid Overload (Injury, poisoning and procedural complications) | 1 (1)
AV Fistula (Injury, poisoning and procedural complications) | 1 (1)
Aortoiliac Dissection (Injury, poisoning and procedural complications) | 1 (1)
Thrombus (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Hemodynamically Unstable (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Tamponade (Injury, poisoning and procedural complications) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Adult Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAVISTAR THERMOCOOL Catheter (N=233)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrioventricular node ablation (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 6 (6)
Arrhythmia - Not Elsewhere Classified (Cardiac disorders) | 6 (7)
Atrial Tachycardia (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 22 (30)
Biventricular assist device placed (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac - Not Elsewhere Classified (Cardiac disorders) | 6 (6)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Cardiac stents (Cardiac disorders) | 4 (4)
Chest Pain - Not Elsewhere Classified (Cardiac disorders) | 3 (3)
Congestive Heart Failure (Cardiac disorders) | 50 (78)
Coronary Artery Disease (Cardiac disorders) | 6 (6)
Endocarditis (Cardiac disorders) | 1 (1)
Heart Block (Cardiac disorders) | 3 (3)
Heart Transplant (Cardiac disorders) | 2 (2)
Implantable Cardioverter Defibrillator maintenance (Cardiac disorders) | 10 (10)
Implantable Cardioverter Defibrillator shock - Not Elsewhere Classified (Cardiac disorders) | 10 (12)
Mitral valve regurgitation (Cardiac disorders) | 2 (3)
Myocardial Infarction (Cardiac disorders) | 5 (5)
Pericardial effusion (Cardiac disorders) | 2 (2)
Pleural Effusion (Cardiac disorders) | 2 (2)
Thrombus (Cardiac disorders) | 4 (4)
Ventricular Tachycardia (Cardiac disorders) | 68 (125)
Abdominal pain - Not Elsewhere Classified (Gastrointestinal disorders) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Esophageal cancer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 3 (3)
Ulcer (Gastrointestinal disorders) | 1 (1)
Chest Pain - Not Elsewhere Classified (General disorders) | 5 (9)
Chest Pain - Non cardiac (General disorders) | 6 (6)
Diabetes (General disorders) | 1 (1)
Elective - Dental (General disorders) | 1 (1)
Fluid overload (General disorders) | 3 (3)
Pain - Not Elsewhere Classified (General disorders) | 1 (1)
Weakness (General disorders) | 3 (3)
Bacteremia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Fever (Infections and infestations) | 2 (2)
Gangrene (Infections and infestations) | 1 (1)
Infection - Not Elsewhere Classified (Infections and infestations) | 2 (2)
Knee infection (Infections and infestations) | 1 (2)
Methicillin-resistant Staphylococcus aureus (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (9)
Prostatitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 7 (7)
Urinary Tract Infections (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 2 (2)
Arteriovenous fistula (Injury, poisoning and procedural complications) | 1 (1)
Cardiac - Not Elsewhere Classified (Injury, poisoning and procedural complications) | 2 (2)
Fracture - Fibula (Injury, poisoning and procedural complications) | 1 (2)
Fracture - hip (Injury, poisoning and procedural complications) | 1 (1)
Fracture - jaw (Injury, poisoning and procedural complications) | 1 (1)
Fracture - pelvis (Injury, poisoning and procedural complications) | 1 (1)
Fracture - rib (Injury, poisoning and procedural complications) | 1 (1)
Fracture - wrist (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 9 (9)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Spider bite (Injury, poisoning and procedural complications) | 1 (1)
Wound - Not Elsewhere Classified (Injury, poisoning and procedural complications) | 1 (1)
Death (Investigations) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bowel Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cysts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (2)
Vertigo (Nervous system disorders) | 1 (1)
Visual disturbance (Nervous system disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (1)
Renal - Not Elsewhere Classified (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 5 (5)
Hematuria (Renal and urinary disorders) | 1 (1)
Kidney stone (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 5 (5)
Revascularization (Vascular disorders) | 1 (2)
Chest Pain - Not Elsewhere Classified (General disorders) | 1 (1)
Transplant - Not Elsewhere Classified (Investigations) | 1 (1)
Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Biosense Webster for additional information.